CLINICAL TRIAL: NCT02662699
Title: Clinical Signs and Symptoms of Anemia in Patients Over 75 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: HUS n° 6247
Record Dates: First submitted 2016-01-07; First posted 2016-01-25 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Anemia
Keywords: Anemia; Hematologic Diseases; Erythrocytes; Hemoglobin; Hemolytic
MeSH Terms: conditions — Anemia; Hematologic Diseases; Hemolysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia is a common pathology in geriatrics. According to the World Health Organization it affects 23.9% of subjects over 60 years in the world, and 8% of patients over 60 years in Europe. A prevalence that increases with the age and twice in individuals over 85 years.

ELIGIBILITY:
Inclusion criteria:

* Adult over 75 years old, male or female

Exclusion criteria:

* Transfusion within 3 months, acute anemia / deglobulisation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Anemic patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Laboratory tests | 1 hour after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ANDRES, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Médecine Interne, diabète et maladies métaboliques - Médicale B, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No